CLINICAL TRIAL: NCT03714451
Title: Investigating the Effect of Onyx Sorghum on Blood Glucose in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Silver Palate Kitchens Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000023930
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: double blinded randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onyx Group (Experimental): Patients with T2DM will receive food products containing onyx sorghum (Onyx Group).
  Interventions: Dietary Supplement: onyx sorghum
- Wheat Flour Group (Active Comparator): Patients with T2DM will receive food products with wheat flour.
  Interventions: Dietary Supplement: whole wheat flour

INTERVENTIONS:
Dietary Supplement: onyx sorghum — The diet intervention will last a total of 28 days. Per the American Heart Association (AHA) and American Diabetes Association (ADA) recommendations, the daily diet plan will consist of 50-55% carbohydrate, 15-20% protein, and 25-30% fat. In the Onyx Group, 25% of carbohydrate will come from the onyx sorghum, and at least three foods per day (including cereals, bread, muffins, pasta, and smoothie boosters) will contain this.
  Arms: Onyx Group
Dietary Supplement: whole wheat flour — Per the American Heart Association (AHA) and American Diabetes Association (ADA) recommendations, the daily diet plan will consist of 50-55% carbohydrate, 15-20% protein, and 25-30% fat.
  Arms: Wheat Flour Group

SUMMARY:
To evaluate the effect of onyx sorghum on blood glucose levels in patients with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
The plan is to study 24 participants with T2DM, who are otherwise healthy. The study will be double-blinded and randomized. Participants will first attend a screening visit (Visit #1) to determine eligibility. Then, eligible participants will be asked to wear a FreeStyle Libre Pro continuous glucose monitor (CGM) for up to 14 days (Visit #2). After this 14-day CGM session, participants will be randomly assigned (1:1) to one of two groups that will receive: 1) food products containing onyx sorghum (Onyx Group) or 2) food products with wheat flour (Control Group). The diet intervention will last a total of 28 days. Participants will have weekly visits to pick up food and bi-weekly blood draws (no more than 20mL at each visit). They will also be asked to wear the CGM throughout the diet intervention and will record their food intake in a daily food diary to confirm that the diet intervention is being followed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-65 years
* A1c < 8.5%
* BMI > 18.5

Exclusion Criteria:

* known malignancy, anemia, kidney disease, and/or liver disease
* untreated thyroid disease
* uncontrolled hypertension
* initiation of any anti-diabetes medications within the last 3 months
* greater than 5% change in weight in the last 3 months
* current or recent steroid use in the last 3 months
* for women: pregnancy or breastfeeding

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in glycemic variability | day 1
  The continuous glucose monitoring (CGM) consists of a sensor that measures glucose levels from the interstitial tissue. Changes in glucose levels from baseline.
Change in glycemic variability | 14 days
  The continuous glucose monitoring (CGM) consists of a sensor that measures glucose levels from the interstitial tissue. Changes in glucose levels from baseline.
Change in glycemic variability | day 28
  The continuous glucose monitoring (CGM) consists of a sensor that measures glucose levels from the interstitial tissue. Changes in glucose levels from baseline.

SECONDARY OUTCOMES:
Changes in weight | day 1
  change in weight from baseline
Changes in weight | day 14
  change in weight from baseline
Changes in weight | day 28
  change in weight from baseline
Changes in BMI | upon screening
  change in BMI from baseline
Changes in BMI | day 1
  change in BMI from baseline
Changes in BMI | day 14
  change in BMI from baseline
Changes in BMI | day 28
  change in BMI from baseline
Change in glucose levels | upon enrollment
  change in blood glucose levels
Change in glucose levels | day 1
  change in blood glucose levels
Change in glucose levels | day 14
  change in blood glucose levels
Change in glucose levels | day 28
  change in blood glucose levels

OTHER OUTCOMES:
Eating behavior | day 1
  measure of food provided and returned
Eating behavior | day 14
  measure of food provided and returned
Eating behavior | day 28
  measure of food provided and returned

CONTACTS AND LOCATIONS:
Overall Officials: Renata Belfort de Aguiar, MD, PhD, Principal Investigator — Yale School of Medicine Department of Endocrinology
Locations (3):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Yale Center for Clinical Investigation, New Haven, Connecticut